CLINICAL TRIAL: NCT03312946
Title: Effect of Vibro-oscillatory Therapy for Improvement of Body Contour and Appearance of Cellulite.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indústria Brasileira Equipamentos Médicos - IBRAMED (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ibramedmodellata
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Body Fat Distribution; Cellulitis
MeSH Terms: conditions — Cellulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment oscillating vibro (Experimental): treatment such as the Modellata electromedical device (Ibramed), in the abdomen, flanks, thigh posterior, inner thigh and buttocks. Being performed twice a week, with a total duration of 50 minutes to the session, being 10 sessions total to end the treatment.
  Interventions: Device: Modellata

INTERVENTIONS:
Device: Modellata — treatment such as the Modellata electromedical device (Ibramed), in the abdomen, flanks, thigh posterior, inner thigh and buttocks.

SUMMARY:
OBJECTIVE: To evaluate the efficacy of vibro-oscillatory therapy through an electromedical equipment in improving body contour and appearance of cellulite.

SUBJECTS AND METHODS: A prospective and comparative longitudinal clinical study will be performed in 30 women with cellulitis. Patients will be submitted to data collection and evaluation and before and after vibration-oscillatory therapy.

HYPOTHESES: Patients are expected to show improvement in body contour and cellulite after vibration-oscillatory therapy.

STATISTICAL ANALYSIS: A descriptive analysis will be done before and after vibration-oscillatory therapy, with frequency tables for categorical and descriptive variables (mean, standard deviation, median, minimum and maximum values) for continuous or numerical variables. In order to compare the main variables between the groups and the collection times, the analysis of variance (ANOVA) for repeated measures will be used. Tukey's test will be used to compare the groups. The significance level adopted for the statistical tests will be 5% or p <0.05.

DETAILED DESCRIPTION:
After approval by the institutional committee of Research Ethics, the subjects will be approached by the researcher responsible on the day of their evaluation, where they completed the registration form, after a brief analysis of the inclusion and exclusion criteria of the present study, the individuals included in the study will be collection of anthropometric data: weight, height, BMI, perimeter of the treated region, assessment of the degree of gynoid lipodystrophy, clinical inspection and photographic study of the treated area, ultrasound examination to assess the thickness of the dermis and hypodermis and the examination with Cutometer ® to assess the viscoelasticity of the skin.

Patients will be divided according to the degree of cellulite they present and will be treated with vibration therapy, such as the Modellata® electromedical equipment (Ibramed- Brazilian Industry of Electronic Equipment), being performed three times a week for two months totaling 16 sessions by a dermato-functional physiotherapist.

Data collection and evaluation will be performed before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female gender, over 18 years of age;
* With body mass index considered eutrophic;
* Cellulite carriers;
* Non smokers;
* That they agree to participate and sign the TCLE.

Exclusion Criteria:

* Male gender;
* Menopausal women;
* Have undergone aesthetic treatment in the gluteal region and thighs in the last 6 months;
* Patients with skin lesions, such as dermatitis and dermatoses;
* Patients with capillary fragility;
* Patients with acute deep vein thrombosis (DVT);
* On or near cancerous lesions;
* Patients with cardiac pacemaker or other implanted electronic device

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-10-13 (Actual); Primary Completion 2017-12-04 (Estimated); Study Completion 2018-02-04 (Estimated)

PRIMARY OUTCOMES:
Improve body contour | 1 hour per session (10 sessions 5 weeks).
  Perimetry, photos, and ultrasound

SECONDARY OUTCOMES:
Improve appearance of cellulite | 1 hour per session (10 sessions 5 weeks).
  perimetry, photos, ultra son, degree of cellulite

CONTACTS AND LOCATIONS:
Locations (1):
- Ibramed - Indústria Brasileira de Equipamentos Médicos, Amparo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided